CLINICAL TRIAL: NCT02795351
Title: The Effect of the Selective PDE5 Inhibitor, Sildenafil, on Aura and Migraine Headache Induction.
Brief Title: Induction of Migraine Aura With Sildenafil
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Christina Kruuse, Consultant neurologist, associate professor, Herlev Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-15008491
Record Dates: First submitted 2016-04-09; First posted 2016-06-10 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Migraine With Aura
MeSH Terms: conditions — Migraine with Aura | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Sildenafil 100 mg single dose
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — Single oral administration of active or placebo one week apart
  Arms: Active
Drug: Placebo
  Arms: Placebo

SUMMARY:
In a double blind placebo-controlled cross-over study the effect of Sildenafil on aura and migraine headache induction is tested in patient with migraine with aura.

ELIGIBILITY:
Inclusion Criteria:

* Migraine with aura
* Minimum of 2 attacks/year

Exclusion Criteria:

* Any other type of headache, except tension-type headache < 4 days per month
* History of cardio- or cerebrovascular diseases
* Hypertension or hypotension
* Any daily intake of medication, including prophylactic migraine treatment, except oral contraceptives
* Pregnancy and lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Aura and migraine like headache | 14 hours
  Induction of aura reported by an aura diary for 14 hours post medication

SECONDARY OUTCOMES:
Markers of endothelial function in blood | 2 hours
Migraine without aura | 14 hours
  Induction of headache resembling usual migraine attacks

CONTACTS AND LOCATIONS:
Overall Officials: Christina Kruuse, MD, DMSc, Principal Investigator — Department of Neurology, Herlev-Gentofte Hospital
Locations (1):
- Department of Neurology, Herlev-Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Butt JH, S Eddelien H, Kruuse C. The headache and aura-inducing effects of sildenafil in patients with migraine with aura. Cephalalgia. 2022 Sep;42(10):984-992. doi: 10.1177/03331024221088998. Epub 2022 Mar 25. PMID 35332812